CLINICAL TRIAL: NCT03762304
Title: The Effect of Household-based Screening on Blood Pressure Changes in South Africa: a Regression Discontinuity Study
Brief Title: The Effect of Household-based Screening on Blood Pressure Changes in South Africa
Status: Completed | Type: Observational
Sponsor: Till Bärnighausen (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor-Investigator, Till Bärnighausen, Alexander von Humboldt University Professor, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Other Study IDs: RDD - BP - South Africa
Record Dates: First submitted 2018-11-30; First posted 2018-12-03 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Hypertension; Blood Pressure
Keywords: Causal inference; Regression discontinuity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: The intervention group consists of individuals with a measured blood pressure just above the hypertensive cut-off of 140 mmHg systolic or 90 mmHg diastolic blood pressure who have never previously been diagnosed as hypertensive and are not taking medication to lower their blood pressure. The exact upper bound on blood pressure will be determined empirically. Individuals in the intervention group were told that that their blood pressure was high, that high blood pressure can lead to life threatening consequences, that blood pressure control can reduce these negative consequences, and that they should seek follow-up care for their blood pressure.
  Interventions: Other: Household blood pressure screening with care encouragement
- Control group: The control group consists of individuals with a measured blood pressure just below the hypertensive cut-off of 140 mmHg systolic and 90 mmHg diastolic blood pressure who have never previously been diagnosed as hypertensive and are not taking medication to lower their blood pressure. The exact lower bound on blood pressure will be determined empirically. These individuals were not given the care encouragement intervention.

INTERVENTIONS:
Other: Household blood pressure screening with care encouragement — During the household survey visit, survey enumerators collected two measurements of the respondent's blood pressure. If either of the measurements exceeded 140 mmHg systolic or 90 mmHg diastolic, enumerators told participants: "Your blood pressure readings are higher than normal. High blood pressure is dangerous because it makes the heart work too hard. High blood pressure increases the risk of heart disease and stroke. High blood pressure can also cause other problems, such as heart failure, kidney disease, and blindness. You can control high blood pressure by taking action." Then the enumerators recommend that an individual seek medical care within 2 months.
  Groups: Intervention group

SUMMARY:
This study will evaluate the effect of household-based screening and care encouragement for blood pressure on subsequent changes in blood pressure. The study uses a quasi-experimental regression discontinuity design with existing population-based secondary data from the 2008, 2010, 2012, 2014, and 2017 waves of the National Income Dynamics Study in South Africa.

DETAILED DESCRIPTION:
Household-based screening and referral to care for blood pressure may improve blood pressure control at the population level in many low- and middle-income countries.

This observational study will use a quasi-experimental regression discontinuity design to evaluate the effect of household-based screening for blood pressure with care encouragement for potentially hypertensive individuals on subsequent changes in blood pressure over time.

Individuals had their blood pressure measured in the household as part of the National Income Dynamics Study data collection. If individuals had a measured blood pressure in the hypertensive zone, they were told that they had elevated blood pressure, that high blood pressure can lead to life threatening consequences, and that they should seek further care. The study exploits the fact that individuals were given this information based on a hard blood pressure cutoff. Therefore, the investigators will evaluate the causal effect of this household-based intervention in the absence of randomization by comparing individuals with a baseline blood pressure just above and below the cut off.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 30
* Valid blood pressure measurements

Exclusion Criteria:

* Prior diagnosis of hypertension
* Currently taking medication for blood pressure
* Measured with a blood pressure above 140 mmHg systolic or 90 mmHg diastolic in a previous wave of data

Min Age: 30 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals will be drawn from the 2008, 2010, 2012, and 2014 waves of the National Income Dynamics Study (NIDS) with the 2017 wave used only for follow-up. The NIDS is a nationally representative, household-based, survey of families and individuals from across South Africa.
Sampling Method: Probability Sample
Enrollment: 3986 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Two-year change in systolic blood pressure | Approximately two years based on the difference between survey waves in the years 2008, 2010, 2012, 2014, and 2017
  For each survey wave, blood pressure is measured at the household by a trained enumerator using an electronic blood pressure device. The enumerators take two separate measurements during the course of the visit with at least three minutes between measurements with individuals in a seated position. The investigators will take the average of the two systolic blood pressure measurements as their main outcome measure.
Nine-year change in systolic blood pressure | Baseline in 2008 and approximately nine years later in 2017.
  For each survey wave, blood pressure is measured at the household by a trained enumerator using an electronic blood pressure device. The enumerators take two separate measurements during the course of the visit with at least three minutes between measurements with individuals in a seated position. The investigators will take the average of the two systolic blood pressure measurements as their main outcome measure.

SECONDARY OUTCOMES:
Health-seeking behavior | Cross-sectionally in 2010, 2012, 2014, and 2018
  Health-care utilization is measured at the household based on respondents' answer to the survey question: "When did you last consult someone about your health?"
Blood pressure treatment | Cross-sectionally in 2010, 2012, 2014, and 2018
  Whether an individual is currently taking treatment to control their blood pressure is measured during the household survey based on the answer to the question: "Are you currently taking medicine for high blood pressure?"

CONTACTS AND LOCATIONS:
Overall Officials: Nikkil Sudharsanan, PhD, Principal Investigator — Research group leader

IPD SHARING:
Plan to Share IPD: Yes
The data are already publicly available at: http://www.nids.uct.ac.za/nids-data/data-access
Time Frame: Data are already available.
URL: http://www.nids.uct.ac.za/nids-data/data-access